CLINICAL TRIAL: NCT01144247
Title: A Phase I Clinical Trial Evaluating Cellular Immunotherapy With Intratumoral Alloreactive Cytotoxic T Lymphocytes and Interleukin-2 for the Treatment of Recurrent Malignant Gliomas or Meningiomas
Brief Title: Cellular Immunotherapy Study for Brain Cancer
Acronym: alloCTL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCLA 07-09-008; R01CA125244 (NIH)
Record Dates: First submitted 2010-06-11; First posted 2010-06-15 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Gliomas; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Mixed Glioma; Glioblastoma Multiforme; Malignant Meningioma
Keywords: Recurrent Grade III or Grade IV Gliomas; anaplastic astrocytoma; anaplastic oligodendroglioma; anaplastic mixed glioma; glioblastoma multiforme; biotherapy; malignant meningioma
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma; Glioblastoma; Meningioma; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- alloreactive CTL arm (Experimental)
  Interventions: Drug: alloreactive CTL

INTERVENTIONS:
Drug: alloreactive CTL — cellular immunotherapy with alloCTL

SUMMARY:
The purpose of this research study to determine if treating recurrent malignant gliomas with another person's (donor) immune system cells known as aCTL cells, will be safe. This study will also try to determine if persons who receive aCTL's are more or less likely to survive their brain tumor than persons who had similar tumors in the past. Approximately 15 patients will be enrolled at UCLA.

ELIGIBILITY:
INCLUSION CRITERIA

To participate in this clinical trial, patients must meet the following eligibility criteria:

1. Subjects must have a histologically proven diagnosis of malignant glioma or meningioma and been treated with prior standard radiation and chemotherapy. There must be evidence of unequivocal progression by MRI.
2. Tumor must be amenable to resection, and surgical resection must be clinically indicated.
3. Age at least 18 years.
4. Karnofsky performance scale score >60.
5. Adequate hematologic function: a) systemic white blood cell count greater than 2 x 103/mm3, b) platelet count greater than 100,000/mm3, c) hematocrit greater than 25%.
6. Adequate renal function, with creatinine less than two times the upper limit.
7. Adequate hepatic function, with SGOT, alkaline phosphatase, and total bilirubin < 2x upper limit of normal.
8. Patients must have an expected survival of at least three months.
9. Patients must not have a history of HTLV, HIV, syphilis by RPR, hepatitis B and C.
10. Patients must sign an informed consent.

EXCLUSION CRITERIA

Patients will be excluded from the trial if the patients:

1. have multifocal tumors, bihemispheric tumors, infratentorial tumors, or non-surgically accessible tumors.
2. have prior tumor resections where the ventricles were extensively breached.
3. are pregnant or breast-feeding women.
4. are females of child-bearing potential unable or unwilling to practice adequate birth control methods.
5. have contraindications for brain MRI scanning (e.g., intra-ocular metal fragments, cerebral aneurysm clips, pacemaker).
6. have concurrent malignancy, excluding curatively treated basal or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix.
7. have concurrent systemic infection.
8. have any clinically significant, uncontrolled medical illness, as determined by the investigators.
9. are unwilling or unable to comply with procedures required in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | 5 years

SECONDARY OUTCOMES:
Maximum tolerated dose | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Hickey MJ, Malone CC, Erickson KL, Jadus MR, Prins RM, Liau LM, Kruse CA. Cellular and vaccine therapeutic approaches for gliomas. J Transl Med. 2010 Oct 14;8:100. doi: 10.1186/1479-5876-8-100. PMID 20946667
- [Background] Hickey MJ, Malone CC, Erickson KE, Gomez GG, Young EL, Liau LM, Prins RM, Kruse CA. Implementing preclinical study findings to protocol design: translational studies with alloreactive CTL for gliomas. Am J Transl Res. 2012;4(1):114-26. Epub 2012 Jan 10. PMID 22347526
- [Result] Kruse CA, Cepeda L, Owens B, Johnson SD, Stears J, Lillehei KO. Treatment of recurrent glioma with intracavitary alloreactive cytotoxic T lymphocytes and interleukin-2. Cancer Immunol Immunother. 1997 Oct;45(2):77-87. doi: 10.1007/s002620050405. PMID 9390198
- [Result] Kruse, C.A., Rubinstein, D. (2001) Cytotoxic T Lymphocytes Reactive to Patient Major Histocompatibility Proteins for Therapy of Recurrent Primary Brain Tumors, in Brain Tumor Immunotherapy, eds. L.M. Liau, D.P. Becker, T.F. Cloughsey, and D. Bigner, Humana Press, pp. 149-170
- See also: Related Info — http://neurosurgery.ucla.edu/default.cfm